CLINICAL TRIAL: NCT05143580
Title: Preoperative Cognitive Therapy Intervention in Reducing Delirium After Cardiac Surgery
Brief Title: Preoperative Intervention to Reduce Delirium After Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CCH-CT-MZ01
Record Dates: First submitted 2021-10-28; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-10

CONDITIONS: Cardiac Surgery
Keywords: Delirium after cardiac surgery; Cognitive therapy; Gamification
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Acceptance conditions: Patients who are expected to undergo traditional thoracotomy or minimally invasive surgery for cardiac surgery, and those who are over 20 years old and have no cognitive impairment before surgery.
  Excluded conditions: patients diagnosed with aortic dissection, over 80 years of age, and previously admitted to the intensive care unit.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Therapy Group (Experimental): * The anesthesiologist will provide the patient with instructions for preoperative anesthesia.
  * The operating room nurses will introduce the operating room environment and surgical care instructions to the patient.
  * Provide a manual for disease health education.
  * Provide post-operative care and environmental imaging materials, explain the importance of intensive care unit routines and related equipment, indwelling pipelines, related nursing staff, post-operative care methods, and provide imaging and health education manuals for explanation.
  * Use gamification to evaluate: pain relief skills, lung expansion skills.
  Interventions: Behavioral: Cognitive therapy
- Routine Care Group (Placebo Comparator): * The anesthesiologist will provide the patient with instructions for preoperative anesthesia.
  * The operating room nurses will introduce the operating room environment and surgical care instructions to the patient.
  * Provide a manual for disease health education.
  Interventions: Behavioral: Routine care

INTERVENTIONS:
Behavioral: Cognitive therapy — * The anesthesiologist will provide the patient with instructions for preoperative anesthesia.
  * The operating room nurses will introduce the operating room environment and surgical care instructions to the patient.
  * Provide a manual for disease health education.
  * Provide post-operative care and environmental imaging materials, explain the importance of intensive care unit routines and related equipment, indwelling pipelines, related nursing staff, post-operative care methods, and provide imaging and health education manuals for explanation.
  * Use gamification to evaluate: pain relief skills, lung expansion skills.
  Arms: Cognitive Therapy Group
Behavioral: Routine care — * The anesthesiologist will provide the patient with instructions for preoperative anesthesia.
  * The operating room nurses will introduce the operating room environment and surgical care instructions to the patient.
  * Provide a manual for disease health education.
  Arms: Routine Care Group

SUMMARY:
This research is designed for experimental quantitative research and is conducted by simple random sampling. Both the control group and the experimental group provided preoperative routine nursing treatment and preoperative medical teaching manuals. The latter adds cognitive therapy and gamification evaluation. Both groups used CAM-ICU to assess the occurrence and duration of postoperative delirium, and DRS-R-98 was used to assess the severity of delirium. After collection, use SPSS 22.0 statistical software package for analysis and processing. The expected result is that the incidence of delirium, the duration of delirium, and the severity of delirium in the experimental group were significantly lower than those in the control group.

DETAILED DESCRIPTION:
This study is an experimental quantitative research design. Both the control group and the experimental group provide routine nursing treatment and preoperative medical teaching manuals before surgery. The latter adds cognitive therapy and gamification evaluation of "Postoperative Care and Environmental Image Data Explanation". The two groups used CAM-ICU to assess the occurrence and duration of delirium after surgery, and DRS-R-98 was used to assess the severity of delirium. From 2021 to 2022, a simple random sampling method is adopted for patients undergoing cardiac surgery in the intensive care unit of a medical center in Central Taiwan, and a lottery is drawn on the first day of each month to determine the belong to which group in the current month. There were 55 persons in each group, and all subjects had no cognitive impairment. After the collected, it was analyzed and processed with SPSS 22.0 statistical package software.

Expected results: The incidence of delirium, the duration of delirium, and the severity of delirium in the experimental group were significantly lower than the control group.

ELIGIBILITY:
Inclusion Criteria:

* Expected to undergo traditional thoracotomy or minimally invasive surgery for cardiac surgery.
* No cognitive impairment before surgery.

Exclusion Criteria:

* Diagnosed with aortic dissection.
* Previously admitted to the intensive care unit.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium | After surgery, the patient was evaluated at 48 hours.
  * First use the Richmond Restlessness and Sedation Scale (RASS) to assess the state of consciousness. RASS is a 10-point scale. +1 to +4 represent different levels of anxiety, 0 points represent alertness and calmness, and -1 to -5 represent different levels of sedation.
  * When the RASS score is between -3 and +4, then evaluate the Confusion Assessment Method for the intensive care unit (CAM-ICU). The CAM-ICU is a four-step assessment method with items on altered mental status or fluctuating course, inattention, and altered level of consciousness or disorganized thinking.
  * If the evaluation result is the following two combinations, the first combination is mental state change, inattention, and consciousness level change; the second combination is mental state change, inattention, and disorganized thinking. This means that the CAM-ICU is positive and delirium has occurred.
Duration of delirium | Completed through delirium, an average of one month.
  - When using the CAM-ICU assessment system, delirium occurs, and the time from the occurrence to the end of the delirium will be recorded.
Severity of delirium | When delirium occurs, assessment is conducted at 9 am every day until the end of delirium, an average of one month.
  * When delirium occurs, use Delirium Rating Scale-Revised-98 (DRS-R-98) to score the severity of delirium symptoms.
  * DRS-R-98 has a total of 16 scoring items, including 13 delirium severity and 3 diagnosis items. The total score is up to 46 points, of which the highest severity is 39 points. The higher the score, the more serious.
  * Clinically, the total score ≥ 18 points or the severity score ≥ 15 points are used.